CLINICAL TRIAL: NCT05465512
Title: Using Radiomics to Predict Neoadjuvant Chemotherapy Efficacy and Postoperative Adjuvant Chemotherapy Benefit in Advanced Gastric Cancer: a Two-center Study
Brief Title: Using Radiomics to Predict Neoadjuvant Chemotherapy Efficacy
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Principal Investigator, Fujian Medical University
Other Study IDs: FMUUH-001
Record Dates: First submitted 2022-07-12; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Gastric Cancer
Keywords: tumor regression grade; radiomics; neoadjuvant chemotherapy; advanced gastric cancer; chemotherapy benefit
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- good response to neoadjuvant chemotherapy (GRNC): Tumor regression grade (TRG) =0 or 1 was defined as a good response to neoadjuvant chemotherapy (GRNC)
  Interventions: Other: response to neoadjuvant chemotherapy
- poor response to neoadjuvant chemotherapy (PRNC): TRG=2 or 3 was defined as a poor response to neoadjuvant chemotherapy (PRNC).
  Interventions: Other: response to neoadjuvant chemotherapy

INTERVENTIONS:
Other: response to neoadjuvant chemotherapy — Tumor regression grade (TRG) =0 or 1 was defined as a good response to neoadjuvant chemotherapy (GRNC), and TRG=2 or 3 was defined as a poor response to neoadjuvant chemotherapy (PRNC).

SUMMARY:
Neoadjuvant chemotherapy (NC) is an important treatment for advanced gastric cancer (AGC). However, tools that effectively predict the efficacy of NC before treatment are lacking. Computed tomography images before and after NC were used to construct a deep learning-based radiomics signature to predict the efficacy of NC, prognoses and postoperative adjuvant chemotherapy benefit.

DETAILED DESCRIPTION:
Background: Neoadjuvant chemotherapy (NC) is an important treatment for advanced gastric cancer (AGC). However, tools that effectively predict the efficacy of NC before treatment are lacking.

Methods: Computed tomography images before and after NC were used to construct a deep learning-based radiomics signature to predict the efficacy of NC, prognoses and postoperative adjuvant chemotherapy benefit. Tumor regression grade (TRG) =0 or 1 was defined as a good response to neoadjuvant chemotherapy (GRNC), and TRG=2 or 3 was defined as a poor response to neoadjuvant chemotherapy (PRNC). 193 patients with AGC from January 2010 to December 2018 in two different China university hospitals were included in this study. The before neoadjuvant chemotherapy imaging scoring system (BNCISS), imaging change scoring system before and after neoadjuvant chemotherapy (ICSS), which were constructed based on computed tomography images before after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Prospective collection and a retrospective analysis of patients seen from January 2010 to December 2018 at Fujian Medical University Union Hospital (FMUUH) and the First Hospital of Lanzhou University (FHLU) who were diagnosed with gastric adenocarcinoma and underwent radical resection

Exclusion Criteria:

* Patients with concurrent malignant disease, distant metastases, palliative resection, or gastric stump cancer were excluded.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Prospective collection and a retrospective analysis of patients seen from January 2010 to December 2018 at Fujian Medical University Union Hospital (FMUUH) and the First Hospital of Lanzhou University (FHLU) who were diagnosed with gastric adenocarcinoma and underwent radical resection yielded 193 neoadjuvant chemotherapy (NC) patients, including 148 cases from FMUUH (derivation cohort) and 45 cases from the FHLU (validation cohort). Of the 148 patients from FMUUH, 139 had computed tomography (CT) images before NC, 141 had CT images after NC, and 132 had CT images before and after NC. All 45 patients in the FHLU underwent CT before and after NC. Patients with concurrent malignant disease, distant metastases, palliative resection, or gastric stump cancer were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
AUC for ICSS | 2022-01-01 to 2022-07-31
  The predictive performance of imaging change scoring system before and after neoadjuvant chemotherapy (ICSS)
AUC for BNCISS | 2022-01-01 to 2022-07-31
  The predictive performance of before neoadjuvant chemotherapy imaging scoring system (BNCISS)

SECONDARY OUTCOMES:
overall survival | 2010-01-01 to 2022-07-31
  3 year overall survival
disease free survival | 2010-01-01 to 2022-07-31
  3 year disease free survival

CONTACTS AND LOCATIONS:
Overall Officials: Hualong Zheng, Study Director — 291167038@qq.com
Locations (1):
- Department of Gastric Surgery, Fuzhou, Fujian, China